CLINICAL TRIAL: NCT01197521
Title: (OSKIRA-1): A Phase III, Multi-centre, Randomised, Double-Blind, Placebo-Controlled, Parallel Group Study of Two Dosing Regimens of Fostamatinib Disodium in Rheumatoid Arthritis Patients With an Inadequate Response to Methotrexate
Brief Title: Evaluation of Effectiveness of Two Dosing Regimens of Fostamatinib Compared to Placebo in Patients With Rheumatoid Arthritis (RA) Who Are Taking Methotrexate But Not Responding.
Acronym: OSKIRA - 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D4300C00001; 2010-020743-12 (EudraCT Number)
Record Dates: First submitted 2010-09-08; First posted 2010-09-09 (Estimated); Results first posted 2014-04-07 (Estimated); Last update posted 2014-04-07 (Estimated); Status verified 2014-02

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — fostamatinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Dosing Regimen A (Experimental): Oral Treatment
  Interventions: Drug: fostamatinib
- Dosing Regimen B (Experimental): Oral Treatment
  Interventions: Drug: fostamatinib
- Dosing Regimen C (Placebo Comparator): Oral Treatment
  Interventions: Drug: placebo, fostamatinib

INTERVENTIONS:
Drug: fostamatinib — fostamatinib 100 mg twice daily
  Arms: Dosing Regimen A
Drug: fostamatinib — fostamatinib 100 mg twice daily/150 mg once daily
  Arms: Dosing Regimen B
Drug: placebo, fostamatinib — Placebo for 24 weeks followed by fostamatinib 100 mg twice daily
  Arms: Dosing Regimen C

SUMMARY:
The purpose of the study is to evaluate the effectiveness of two dosing regimens of fostamatinib compared to placebo, in patients with rheumatoid arthritis (RA) who are taking methotrexate but not responding. The study will last for 1 year.

DETAILED DESCRIPTION:
Sub-study:

Full title: Optional Genetic Research

Date: 18 June 2010

Version: 1

Objectives: To collect and store, with appropriate consent ,DNA samples for future exploratory research into genes/genetic variation that may influence response (ie, absorption, distribution, metabolism and excretion, safety, tolerability and efficacy) to fostamatinib disodium and/or methotrexate; and/or susceptibility to, progression of and prognosis of RA

ELIGIBILITY:
Inclusion Criteria:

* Active rheumatoid arthritis (RA) diagnosed after the age of 16
* Currently taking methotrexate
* 6 or more swollen joints and 6 or more tender/painful joints (from 28 joint count) and either Erythrocyte Sedimentation Rate (ESR) blood result of 28mm/h or more, or C-Reactive Protein (CRP) blood result of 10mg/L or more
* At least one of the following: documented history of positive rheumatoid factor (blood test), current presence of rheumatoid factor (blood test), radiographic erosion within 12 months prior to study enrolment, presence of serum anti-cyclic citrullinated peptide antibodies (blood test)

Exclusion Criteria:

* Females who are pregnant or breast feeding
* Poorly controlled hypertension
* Liver disease or significant liver function test abnormalities
* Certain inflammatory conditions (other than rheumatoid arthritis), connective tissue diseases or chronic pain disorders
* Recent or significant cardiovascular disease
* Significant active or recent infection including tuberculosis
* Previous failure to respond to a TNF alpha antagonist, anakinra or previous treatment with other biological agent
* Severe renal impairment
* Neutropenia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 923 (Actual)
Dates: Start 2010-09; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neil MacKillop, MD PhD, Study Director — AstraZeneca
Locations (127):
- United States (41):
  - Research Site, Anniston, Alabama
  - Research Site, Huntsville, Alabama
  - Research Site, Tuscaloosa, Alabama
  - Research Site, Tucson, Arizona
  - Research Site, Huntington Beach, California
  - Research Site, Long Beach, California
  - Research Site, Santa Maria, California
  - Research Site, Santa Monica, California
  - Research Site, Colorado Springs, Colorado
  - Research Site, Bridgeport, Connecticut
  - Research Site, Lewes, Delaware
  - Research Site, Daytona Beach, Florida
  - Research Site, Ocala, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Marietta, Georgia
  - Research Site, Idaho Falls, Idaho
  - Research Site, Springfield, Illinois
  - Research Site, Wichita, Kansas
  - Research Site, Bowling Green, Kentucky
  - Research Site, Flowood, Mississippi
  - Research Site, Florissant, Missouri
  - Research Site, Richmond Heights, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Kalispell, Montana
  - Research Site, Albuquerque, New Mexico
  - Research Site, Albany, New York
  - Research Site, Brooklyn, New York
  - Research Site, Olean, New York
  - Research Site, Asheville, North Carolina
  - Research Site, Greensboro, North Carolina
  - Research Site, Perrysburg, Ohio
  - Research Site, Lake Oswego, Oregon
  - Research Site, Erie, Pennsylvania
  - Research Site, Waxford, Pennsylvania
  - Research Site, Charleston, South Carolina
  - Research Site, Hixson, Tennessee
  - Research Site, Memphis, Tennessee
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, Mesquite, Texas
  - Research Site, San Antonio, Texas
- Argentina (9):
  - Research Site, Reading, Berkshire
  - Research Site, Buenos Aires, Buenos Aires F.D.
  - Research Site, Ciudad Autonoma Bs As, CBA
  - Research Site, Córdoba, CRD
  - Research Site, San Juan, San Juan Province
  - Research Site, Rosario, Santa Fe Province
  - Research Site, San Miguel de Tucumán, TUC
  - Research Site, Caba
  - Research Site, Quilmes
- Australia (3):
  - Research Site, Camperdown, New South Wales
  - Research Site, Cairns, Queensland
  - Research Site, Southport, Queensland
- Belgium (2):
  - Research Site, Brussels
  - Research Site, Yvoir
- Brazil (5):
  - Research Site, Vitória, Espírito Santo
  - Research Site, Curitiba, Paraná
  - Research Site, Recife, Pernambuco
  - Research Site, São Paulo, São Paulo
  - Research Site, Rio de Janeiro
- Bulgaria (4):
  - Research Site, Plovdiv
  - Research Site, Sevlievo
  - Research Site, Sofia
  - Research Site, Veliko Tarnovo
- Chile (2):
  - Research Site, Osorno, Los Lagos Region
  - Research Site, Santiago
- Estonia (3):
  - Research Site, Pärnu
  - Research Site, Tallinn
  - Research Site, Tartu
- France (2):
  - Research Site, Orléans
  - Research Site, Paris
- Hungary (8):
  - Research Site, Balatonfüred
  - Research Site, Békéscsaba
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Makó
  - Research Site, Sopron
  - Research Site, Szentes
  - Research Site, Zalaegerszeg-pozva
- India (10):
  - Research Site, Secunderabad, Andhra Pradesh
  - Research Site, Visakhapatnam, Andhra Pradesh
  - Research Site, Ahmedabad, Gujarat
  - Research Site, Bangalore, Karnataka
  - Research Site, Mangalore, Karnataka
  - Research Site, Udupi, Karnataka
  - Research Site, Nagpur, Maharshtra
  - Research Site, Lucknow, Uttar Pradesh
  - Research Site, Hyderabad
  - Research Site, Kolkata
- Mexico (8):
  - Research Site, Chihuahua City, Chihuahua
  - Research Site, Saltillo, Coahuila
  - Research Site, Guadalajara, Jalisco
  - Research Site, Mexico City, Mexico City
  - Research Site, San Luis Potosi, Mexico
  - Research Site, Monterrey, Nuevo León
  - Research Site, Obrergon, Sonora
  - Research Site, Mexicali
- Peru (3):
  - Research Site, Arequipa, Arequipa
  - Research Site, Lima, Lima Province
  - Research Site, Pueblo Libre, Lima region
- Poland (8):
  - Research Site, Bytom
  - Research Site, Chełm Śląski
  - Research Site, Grodzisk Mazowiecki
  - Research Site, Katowice
  - Research Site, Krakow
  - Research Site, Warsaw
  - Research Site, Wroclaw
  - Research Site, Żyrardów
- Slovakia (4):
  - Research Site, Bratislava, Slovakia
  - Research Site, Žilina, Slovakia
  - Research Site, Poprad
  - Research Site, Rimavská Sobota
- Ukraine (9):
  - Research Site, Donetsk
  - Research Site, Ivano-Frankivsk
  - Research Site, Kharkiv
  - Research Site, Kiev
  - Research Site, Kyiv
  - Research Site, Lviv
  - Research Site, Odesa
  - Research Site, Vinnytsia
  - Research Site, Zaporyzhzhya
- United Kingdom (6):
  - Research Site, Warrington, Cheshire
  - Research Site, Christchurch
  - Research Site, Ipswich
  - Research Site, London
  - Research Site, Metropolitan Borough of Wirral
  - Research Site, Westcliff-on-the Sea

REFERENCES:
- [Derived] Kjelgaard-Petersen CF, Platt A, Braddock M, Jenkins MA, Musa K, Graham E, Gantzel T, Slynn G, Weinblatt ME, Karsdal MA, Thudium CS, Bay-Jensen AC. Translational Biomarkers and Ex Vivo Models of Joint Tissues as a Tool for Drug Development in Rheumatoid Arthritis. Arthritis Rheumatol. 2018 Sep;70(9):1419-1428. doi: 10.1002/art.40527. Epub 2018 Jul 24. PMID 29669391

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 1475 patients were enrolled: 311, 306 & 306 were randomised to Groups A, B & C, respectively (310, 304 & 304 received at least 1 dose of IP).
Pre-assignment Details: A total of 552 patients failed screening.
Groups:
- FOSTA 100 MG BID PO: Dosing Group A
- FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO: Dosing Group B
- PLACEBO (24 WKS) THEN FOSTA 100 MG BID PO: Dosing Group C
Period: Overall Study
Arm/Group | FOSTA 100 MG BID PO | FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO | PLACEBO (24 WKS) THEN FOSTA 100 MG BID PO
Started | 310 (Patients who received treatment) | 304 (Patients who received treatment) | 304 (Patients who received treatment)
Randomised But Did Not Receive Treatment | 1 (Eligibility criteria not fulfilled) | 2 (Eligibility criteria not fulfilled/other) | 2 (Adverse event/eligibility criteria not fulfilled)
Completed | 207 (Number of patients who completed treatment includes patients who had a dose reduction.) | 191 (Number of patients who completed treatment includes patients who had a dose reduction.) | 161 (Number of patients who completed treatment includes patients who had a dose reduction.)
Not Completed | 103 | 113 | 143
Not completed — Not reported | 24 | 25 | 21
Not completed — Enrolment in long term extension | 42 | 36 | 87
Not completed — Severe non-compliance to protocol | 1 | 3 | 3
Not completed — Lack of therapeutic response | 2 | 3 | 4
Not completed — Dev. of study specific discont. criteria | 6 | 16 | 2
Not completed — Lost to Follow-up | 3 | 2 | 2
Not completed — Adverse Event | 25 | 28 | 24

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FOSTA 100 MG BID PO | FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO | PLACEBO (24 WKS) THEN FOSTA 100 MG BID PO | Total
Number analyzed (Participants) | 310 | 304 | 304 | 918
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (12.2) | 52 (12.0) | 53 (11.9) | 52 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 263 | 254 | 253 | 770
  Male | 47 | 50 | 51 | 148
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 218 | 213 | 209 | 640
  Black or African American | 9 | 5 | 11 | 25
  Asian | 3 | 10 | 5 | 18
  American Indian or Alaska Native | 14 | 12 | 11 | 37
  Indian or Pakistani | 20 | 14 | 19 | 53
  Other | 46 | 50 | 49 | 145

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With ACR20 at Week 24, Comparison Between Fostamatinib and Placebo.
Description: ACR20: American College of Rheumatology 20% response criteria, based on count of swollen and tender joints (out of 28 joints), blood test measures of inflammation (such as CRP) and the physician and patient's own assessments of disease activity, pain and physical function. Non-responder imputation has been applied by carrying the baseline observation forward. BID=twice daily, CRP=C-reactive protein, DMARD=disease-modifying anti-rheumatic drug, PO=orally, QD=once a day.
Time Frame: 24 weeks
Population: The full analysis set includes those patients who received at least 1 dose of investigational product. Patients were analysed by randomised treatment in accordance with the intention to treat principle.
Measure: Number; unit: Percentage of responders
Arm/Group | FOSTA 100 MG BID PO | FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO | PLACEBO (24 WKS) THEN FOSTA 100 MG BID PO
Number analyzed (Participants) | 310 | 304 | 304
Percentage of responders | 49.0 | 44.4 | 34.2
Statistical Analysis 1: Comparison: FOSTA 100 MG BID PO vs PLACEBO (24 WKS) THEN FOSTA 100 MG BID PO; Non-responder imputation has been applied following premature withdrawal, or increased dose of methotrexate or any DMARD initiation, or for 8 weeks following receipt of any parenteral steroids, or for patients with no post baseline data; Test type: Superiority or Other; p < 0.001, Mantel Haenszel — Week 24; Treatment difference in proportion of responders with a Mantel Haenszel approach stratified by pooled country; Weighted difference in proportions = 0.15, 95% CI 2-sided [0.08 to 0.22]
Statistical Analysis 2: Comparison: FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO vs PLACEBO (24 WKS) THEN FOSTA 100 MG BID PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.006, Mantel Haenszel — Week 24; Treatment difference in proportion of responders with a Mantel Haenszel approach stratified by pooled country; Weighted difference in proportions = 0.10, 95% CI 2-sided [0.03 to 0.18]

2. Primary Outcome: Change From Baseline to Week 24 in mTSS, Comparison Between Fostamatinib and Placebo.
Description: mTSS: modified total Sharp score, a measure of structural progression based upon X-rays. Hand and foot joints are scored for erosions and joint space narrowing and the results summed to give a value between 0 and 448. A higher value represents more serious progression of the disease. After disregarding ineligible records, patients with 2 or more non-missing values have had missing data imputed via linear extrapolation/interpolation methods. Patients with only 1 result have been excluded from the analysis. ANCOVA=analysis of covariance, BID=twice daily, DMARD=disease-modifying anti-rheumatic drug, IP=investigational product, PO=orally, QD=once a day.
Time Frame: Baseline and 24 weeks
Population: The full analysis set includes those patients who received at least 1 dose of IP. Patients were analysed by randomised treatment. Measurements at 2 timepoints are required in order for a patient to be included in the analysis; therefore patients with only 1 result have been excluded from the analysis population.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | FOSTA 100 MG BID PO | FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO | PLACEBO (24 WKS) THEN FOSTA 100 MG BID PO
Number analyzed (Participants) | 285 | 277 | 278
Units on a scale | 0.45 (2.201) | 1.29 (13.380) | 0.13 (2.142)
Statistical Analysis 1: Comparison: FOSTA 100 MG BID PO vs PLACEBO (24 WKS) THEN FOSTA 100 MG BID PO; This analysis is performed using an ANCOVA model on the ranks of the change from baseline, by pooled country, including a term for the ranks of the baseline score as a covariate; Test type: Superiority or Other; p = 0.252, Cochran-Mantel-Haenszel — Week 24; The residuals from the ANCOVA are analysed using a Cochran-Mantel-Haenszel approach, adjusting for the effects of pooled country
Statistical Analysis 2: Comparison: FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO vs PLACEBO (24 WKS) THEN FOSTA 100 MG BID PO; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.170, Cochran-Mantel-Haenszel — Week 24; [statistical method as in outcome 2, analysis 1]

3. Secondary Outcome: ACR20 - Proportion of Patients Achieving ACR20, Comparison Between Fostamatinib and Placebo at Week 1
Description: ACR20: American College of Rheumatology 20% response criteria, based on count of swollen and tender joints (out of 28 joints), blood test measures of inflammation (such as CRP) and the physician and patient's own assessments of disease activity, pain and physical function. Non-responder imputation has been applied by carrying the baseline observation forward. BID=twice daily, CRP=C-reactive protein, DMARD=Disease-modifying anti-rheumatic drug, PO=orally.
Time Frame: 1 week
Population: as for outcome 1
Measure: Number; unit: Percentage of responders
Groups:
- FOSTA 100 MG BID (Combined): Dosing Group A and B combined
Arm/Group | FOSTA 100 MG BID (Combined) | PLACEBO (24 WKS) THEN FOSTA 100 MG BID PO
Number analyzed (Participants) | 614 | 304
Percentage of responders | 18.2 | 4.9
Statistical Analysis 1: Comparison: FOSTA 100 MG BID (Combined) vs PLACEBO (24 WKS) THEN FOSTA 100 MG BID PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Mantel Haenszel — Nominal p-values presented. Formal statistical testing could not be carried out due to the predefined multiplicity procedure (as the primary variable comparisons were non-significant); 95% confidence intervals and p-values are calculated using a Mantel Haenszel approach stratified by pooled country; Weighted difference in proportion = 0.13, 95% CI 2-sided [0.10 to 0.17]

4. Secondary Outcome: Proportion of Patients Achieving ACR50 up to Week 24
Description: ACR50: American College of Rheumatology 50% response criteria, based on count of swollen and tender joints (out of 28 joints), blood test measures of inflammation (such as CRP) and the physician and patient's own assessments of disease activity, pain and physical function. Non-responder imputation has been applied by carrying the baseline observation forward. BID=twice daily, CRP=C-reactive protein, DMARD=Disease-modifying anti-rheumatic drug, PO=orally, QD=once a day.
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of responders
Arm/Group | FOSTA 100 MG BID PO | FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO | PLACEBO (24 WKS) THEN FOSTA 100 MG BID PO
Number analyzed (Participants) | 310 | 304 | 304
Percentage of responders | 26.1 | 18.4 | 9.9
Statistical Analysis 1: Comparison: FOSTA 100 MG BID PO vs PLACEBO (24 WKS) THEN FOSTA 100 MG BID PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Mantel Haenszel — [p-value comment as in outcome 3, analysis 1]; 95% confidence intervals and p-values are calculated using a Mantel Haenszel approach stratified by pooled country; Weighted difference in proportions = 0.16, 95% CI 2-sided [0.11 to 0.22]
Statistical Analysis 2: Comparison: FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO vs PLACEBO (24 WKS) THEN FOSTA 100 MG BID PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.002, Mantel Haenszel — [p-value comment as in outcome 3, analysis 1]; 95% confidence intervals and p-values are calculated using a Mantel Haenszel approach stratified by pooled country; Weighted difference in proportions = 0.09, 95% CI 2-sided [0.03 to 0.14]

5. Secondary Outcome: Proportion of Patients Achieving ACR70 up to Week 24
Description: ACR70: American College of Rheumatology 70% response criteria, based on count of swollen and tender joints (out of 28 joints), blood test measures of inflammation (such as CRP) and the physician and patient's own assessments of disease activity, pain and physical function. Non-responder imputation has been applied by carrying the baseline observation forward. BID=twice daily, CRP=C-reactive protein, DMARD=Disease-modifying anti-rheumatic drug, PO=orally, QD=once a day.
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of responders
Arm/Group | FOSTA 100 MG BID PO | FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO | PLACEBO (24 WKS) THEN FOSTA 100 MG BID PO
Number analyzed (Participants) | 310 | 304 | 304
Percentage of responders | 10.3 | 5.6 | 2.0
Statistical Analysis 1: Comparison: FOSTA 100 MG BID PO vs PLACEBO (24 WKS) THEN FOSTA 100 MG BID PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Mantel Haenszel — [p-value comment as in outcome 3, analysis 1]; 95% confidence intervals and p-values are calculated using a Mantel Haenszel approach stratified by pooled country; Weighted difference in proportions = 0.08, 95% CI 2-sided [0.05 to 0.12]
Statistical Analysis 2: Comparison: FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO vs PLACEBO (24 WKS) THEN FOSTA 100 MG BID PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.015, Mantel Haenszel — [p-value comment as in outcome 3, analysis 1]; 95% confidence intervals and p-values are calculated using a Mantel Haenszel approach stratified by pooled country; Weighted difference in proportions = 0.04, 95% CI 2-sided [0.01 to 0.07]

6. Secondary Outcome: ACRn - Comparison Between Fostamatinib and Placebo at Week 24
Description: ACRn: American College of Rheumatology index of RA improvement, based on smallest percentage improvement in the count of swollen joints (out of 28 joints), count of tender joints (out of 28 joints), or in blood test measures of inflammation (such as CRP) or the physician or patient's own assessments of disease activity, pain and physical function. Scores are reported as a percentage improvement on a scale of -100 to +100, with larger values representing a better clinical outcome. BID=twice daily, CI=confidence interval, CRP=C-reactive protein, DMARD=Disease-modifying anti-rheumatic drug, PO=orally, QD=once a day, RA=rheumatoid arthritis. Mean refers to change at Week 24.
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage improvement from baseline
Arm/Group | FOSTA 100 MG BID PO | FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO | PLACEBO (24 WKS) THEN FOSTA 100 MG BID PO
Number analyzed (Participants) | 310 | 304 | 304
Percentage improvement from baseline | 26.13 (30.833) | 20.06 (28.599) | 12.92 (26.611)
Statistical Analysis 1: Comparison: FOSTA 100 MG BID PO vs PLACEBO (24 WKS) THEN FOSTA 100 MG BID PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Van Elteren — Nominal p-value presented for treatment comparison. ACRn was not formally tested within the predefined multiplicity procedure. As this is a non-parametric test p-values alone are presented rather than an estimated treatment difference; The treatment differences, 95% CIs and p-values are estimated using the Van Elteren test stratified by pooled country
Statistical Analysis 2: Comparison: FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO vs PLACEBO (24 WKS) THEN FOSTA 100 MG BID PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.002, Van Elteren — [p-value comment as in outcome 6, analysis 1]; The treatment differences, 95% CIs and p-values are estimated using the Van Elteren test stratified by pooled country

7. Secondary Outcome: Proportion of Patients Achieving DAS28-CRP <2.6 at Week 12
Description: DAS28-CRP: Disease Activity Score based on a count of swollen and tender joints (out of 28 joints), blood test measures of inflammation (CRP) and the patient's own assessment. Scores can take any positive value with a lower value indicating a better clinical condition. A DAS28-CRP score of <2.6 is indicative of remission of RA symptoms. BID=twice daily, CRP=C-reactive protein, DMARD=Disease-modifying anti-rheumatic drug, OR=odds ratio, PO=orally, QD=once a day.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of responders
Arm/Group | FOSTA 100 MG BID PO | FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO | PLACEBO (24 WKS) THEN FOSTA 100 MG BID PO
Number analyzed (Participants) | 310 | 304 | 304
Percentage of responders | 10.3 | 7.9 | 2.0
Statistical Analysis 1: Comparison: FOSTA 100 MG BID PO vs PLACEBO (24 WKS) THEN FOSTA 100 MG BID PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Regression, Logistic — [p-value comment as in outcome 3, analysis 1]; Odds ratio and 95% confidence intervals are calculated using Logistic Regression with treatment and pooled country as factors; Odds Ratio (OR) = 6.0, 95% CI 2-sided [2.44 to 14.64] — An odds ratio >1 indicates a benefit towards Fostamatinib
Statistical Analysis 2: Comparison: FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO vs PLACEBO (24 WKS) THEN FOSTA 100 MG BID PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.002, Regression, Logistic — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 7, analysis 1]; Odds Ratio (OR) = 4.4, 95% CI 2-sided [1.76 to 11.02] — An odds ratio >1 indicates a benefit towards Fostamatinib

8. Secondary Outcome: Proportion of Patients Achieving DAS28-CRP <2.6 at Week 24
Description: as for outcome 7
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of responders
Arm/Group | FOSTA 100 MG BID PO | FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO | PLACEBO (24 WKS) THEN FOSTA 100 MG BID PO
Number analyzed (Participants) | 310 | 304 | 304
Percentage of responders | 13.2 | 8.6 | 4.9
Statistical Analysis 1: Comparison: FOSTA 100 MG BID PO vs PLACEBO (24 WKS) THEN FOSTA 100 MG BID PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Regression, Logistic — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 7, analysis 1]; Odds Ratio (OR) = 3.0, 95% CI 2-sided [1.63 to 5.67] — An odds ratio >1 indicates a benefit towards Fostamatinib
Statistical Analysis 2: Comparison: FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO vs PLACEBO (24 WKS) THEN FOSTA 100 MG BID PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.083, Regression, Logistic — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 7, analysis 1]; Odds Ratio (OR) = 1.8, 95% CI 2-sided [0.93 to 3.50] — An odds ratio >1 indicates a benefit towards Fostamatinib

9. Secondary Outcome: Proportion of Patients Achieving DAS28-CRP EULAR Response at Week 24
Description: Change in DAS28 was derived for each post baseline scheduled assessment and categorised using the European League Against Rheumatism (EULAR) response criteria. Non-responder imputation has been applied by carrying the baseline observation forward. BID=twice daily, CRP=C-reactive protein, DAS28=Disease Activity Score based on a 28-joint count, DMARD=disease-modifying anti-rheumatic drug, OR=odds ratio, PO=orally, QD=once a day.
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of responders
Arm/Group | FOSTA 100 MG BID PO | FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO | PLACEBO (24 WKS) THEN FOSTA 100 MG BID PO
Number analyzed (Participants) | 310 | 304 | 304
Percentage of responders
  No response | 34.8 (1.46) [0.20 to 0.68] | 41.1 (1.34) [0.26 to 0.89] | 53.0 (1.30) [0.20 to 0.65]
  Moderate response | 39.0 | 44.4 | 36.2
  Good response | 26.1 | 14.5 | 10.9
Statistical Analysis 1: Comparison: FOSTA 100 MG BID PO vs PLACEBO (24 WKS) THEN FOSTA 100 MG BID PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Proportional odds model — Nominal p-value presented for treatment comparison. This was not formally tested within the predefined multiplicity procedure; No response, moderate response and good response are included in the proportional odds model with treatment and pooled country as factors; Odds Ratio (OR) = 2.43, 95% CI 2-sided [1.79 to 3.30] — An odds ratio >1 indicates a benefit towards fostamatinib
Statistical Analysis 2: Comparison: FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO vs PLACEBO (24 WKS) THEN FOSTA 100 MG BID PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.004, Proportional odds model — [p-value comment as in outcome 9, analysis 1]; [statistical method as in outcome 9, analysis 1]; Odds Ratio (OR) = 1.57, 95% CI 2-sided [1.16 to 2.14] — An odds ratio >1 indicates a benefit towards Fostamatinib

10. Secondary Outcome: HAQ-DI Response - Comparison of the Change (>=0.22) From Baseline Between Fostamatinib and Placebo at Week 24
Description: HAQ-DI: Health Assessment Questionnaire - Disability Index, a measure of physical function. The HAQ-DI score is calculated by summing scores from 8 sub-categories (ie, scores for patient ability in dressing and grooming, rising, eating, walking, hygiene, reach, grip and common daily activities) and dividing by the number of categories completed. The HAQ-DI score takes values between 0 and 3, with higher score indicating greater disability. HAQ-DI response: a reduction from baseline in HAQ-DI greater than or equal to the minimally important difference (0.22). BID=twice daily, DMARD=disease-modifying anti-rheumatic drug, OR=odds ratio, PO=orally, QD=once a day.
Time Frame: Baseline and 24 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of responders
Arm/Group | FOSTA 100 MG BID PO | FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO | PLACEBO (24 WKS) THEN FOSTA 100 MG BID PO
Number analyzed (Participants) | 310 | 304 | 304
Percentage of responders | 54.8 | 50.3 | 35.2
Statistical Analysis 1: Comparison: FOSTA 100 MG BID PO vs PLACEBO (24 WKS) THEN FOSTA 100 MG BID PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Regression, Logistic — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 7, analysis 1]; Odds Ratio (OR) = 2.3, 95% CI 2-sided [1.68 to 3.26] — An odds ratio >1 indicates a benefit towards Fostamatinib
Statistical Analysis 2: Comparison: FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO vs PLACEBO (24 WKS) THEN FOSTA 100 MG BID PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Regression, Logistic — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 7, analysis 1]; Odds Ratio (OR) = 1.9, 95% CI 2-sided [1.38 to 2.68] — An odds ratio >1 indicates a benefit towards Fostamatinib

11. Secondary Outcome: SF-36 - Comparison of the Change in PCS From Baseline Between Fostamatinib and Placebo at Week 24
Description: SF-36: 36 item Short Form Health Survey, a measure of health-related QoL. Scores for 8 sub-domains (Physical Functioning, Role-physical, Bodily Pain, General Health, Vitality, Social Function, Role-emotional & Mental Health) are derived & normalised to a scale of 0-100. Physical Component Scores (PCS) are derived by multiplying each of these 8 scores by a constant, summing them & standardising against a population with mean of 50, standard deviation of 10. Higher scores represent a better QoL. Mean changes from baseline score are presented at each visit as increases from baseline (defined as post-baseline minus baseline); larger changes indicate a better clinical condition. ANCOVA=analysis of covariance, BID=twice daily, DMARD=disease modifying antirheumatic drug, PO=orally, QD=once daily, QoL=quality of life.
Time Frame: Baseline and 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | FOSTA 100 MG BID PO | FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO | PLACEBO (24 WKS) THEN FOSTA 100 MG BID PO
Number analyzed (Participants) | 310 | 304 | 303
Units on a scale | 6 (8.0) | 5 (6.7) | 3 (6.2)
Statistical Analysis 1: Comparison: FOSTA 100 MG BID PO vs PLACEBO (24 WKS) THEN FOSTA 100 MG BID PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 9, analysis 1]; Including terms for baseline as a continuous covariate and treatment and pooled country as factors; Treatment difference = 2.24, 95% CI [1.16 to 3.31]
Statistical Analysis 2: Comparison: FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO vs PLACEBO (24 WKS) THEN FOSTA 100 MG BID PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.020, ANCOVA — [p-value comment as in outcome 9, analysis 1]; Including terms for baseline as a continuous covariate and treatment and pooled country as factors; Treatment difference = 1.27, 95% CI [0.20 to 2.35]

12. Secondary Outcome: SF-36 - Comparison of the Change in MCS From Baseline Between Fostamatinib and Placebo at Week 24
Description: SF-36: 36 item Short Form Health Survey, a measure of health-related QoL. Scores for 8 sub-domains (Physical Functioning, Role-physical, Bodily Pain, General Health, Vitality, Social Function, Role-emotional & Mental Health) are derived & normalised to a scale of 0-100. Mental Component Scores (MCS) are derived by multiplying each of these 8 scores by a constant, summing them & standardising against a population with mean of 50, standard deviation of 10. Higher scores represent a better QoL. Mean changes from baseline score are presented at each visit as increases from baseline (defined as post-baseline minus baseline); larger changes indicate a better clinical condition. ANCOVA=analysis of covariance, BID=twice daily, DMARD=disease modifying antirheumatic drug, PO=orally, QD=once daily, QoL=quality of life.
Time Frame: Baseline and 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | FOSTA 100 MG BID PO | FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO | PLACEBO (24 WKS) THEN FOSTA 100 MG BID PO
Number analyzed (Participants) | 310 | 304 | 303
Units on a scale | 4 (9.5) | 4 (8.6) | 2 (8.1)
Statistical Analysis 1: Comparison: FOSTA 100 MG BID PO vs PLACEBO (24 WKS) THEN FOSTA 100 MG BID PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.005, ANCOVA — [p-value comment as in outcome 9, analysis 1]; Including terms for baseline as a continuous covariate and treatment and pooled country as factors; Treatment difference = 1.80, 95% CI [0.54 to 3.07]
Statistical Analysis 2: Comparison: FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO vs PLACEBO (24 WKS) THEN FOSTA 100 MG BID PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.017, ANCOVA — [p-value comment as in outcome 9, analysis 1]; Including terms for baseline as a continuous covariate and treatment and pooled country as factors; Treatment difference = 1.56, 95% CI [0.28 to 2.83]

ADVERSE EVENTS:
Time Frame: 52 weeks
Description: For placebo treated patients time frame includes both placebo (24 weeks) and fostamatinib (28 weeks) treatment. 5 SAEs occurred during the 24 week placebo treated period.
Groups:
- FOSTA 100 MG BID: Dosing Group A
- FOSTA 100 MG BID (4 WKS) THEN 150 MG QD: Dosing Group B
- PLACEBO (24 WKS) THEN FOSTA 100 MG BID - FOSTA Period: Dosing Group C
Arm/Group | FOSTA 100 MG BID | FOSTA 100 MG BID (4 WKS) THEN 150 MG QD | PLACEBO (24 WKS) THEN FOSTA 100 MG BID - FOSTA Period | PLACEBO (24 WKS) THEN FOSTA 100 MG BID - Placebo Period
Serious Adverse Events (participants affected / at risk) | 24/310 | 24/304 | 12/304 | 5/304
Other Adverse Events (participants affected / at risk) | 169/310 | 191/304 | 64/304 | 80/304
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FOSTA 100 MG BID (N=310) | FOSTA 100 MG BID (4 WKS) THEN 150 MG QD (N=304) | PLACEBO (24 WKS) THEN FOSTA 100 MG BID - FOSTA Period (N=304) | PLACEBO (24 WKS) THEN FOSTA 100 MG BID - Placebo Period (N=304)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
ATRIAL FLUTTER (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CARDIAC FAILURE (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CARDIAC FAILURE ACUTE (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CARDIOPULMONARY FAILURE (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CHORIORETINOPATHY (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COLITIS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COLONIC OBSTRUCTION (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DUODENAL ULCER HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ATRIAL THROMBOSIS (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
GASTRITIS ATROPHIC (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PANCREATITIS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
REFLUX GASTRITIS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BILE DUCT OBSTRUCTION (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BILIARY COLIC (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CHOLECYSTITIS (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
CHOLELITHIASIS (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
ANAPHYLACTIC REACTION (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
APPENDICITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BACTERIAL DIARRHOEA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BRONCHITIS (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
CELLULITIS (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
ESCHERICHIA URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
GASTROENTERITIS VIRAL (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PANCREATITIS VIRAL (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PULMONARY TUBERCULOSIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SEPSIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SEPTIC SHOCK (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ACCIDENTAL OVERDOSE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CONTUSION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
FIBULA FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HIP FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SPINAL FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
TIBIA FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
FOOT DEFORMITY (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
PATHOLOGICAL FRACTURE (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
SPONDYLOLISTHESIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SYSTEMIC LUPUS ERYTHEMATOSUS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
GANGLIONEUROMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
GASTRIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
RENAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
THYROID CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
UTERINE LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ISCHAEMIC STROKE (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MULTIPLE SCLEROSIS (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
TRANSIENT GLOBAL AMNESIA (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ABORTION SPONTANEOUS (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CONFUSIONAL STATE (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CALCULUS URINARY (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NEPHROLITHIASIS (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RENAL ARTERY STENOSIS (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
RENAL FAILURE ACUTE (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
HAEMORRHAGIC OVARIAN CYST (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
METRORRHAGIA (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ANGIOEDEMA (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
VITILIGO (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CIRCULATORY COLLAPSE (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPOTENSION (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HYPOVOLAEMIC SHOCK (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PERIPHERAL ISCHAEMIA (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FOSTA 100 MG BID (N=310) | FOSTA 100 MG BID (4 WKS) THEN 150 MG QD (N=304) | PLACEBO (24 WKS) THEN FOSTA 100 MG BID - FOSTA Period (N=304) | PLACEBO (24 WKS) THEN FOSTA 100 MG BID - Placebo Period (N=304)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 12 (12) | 16 (17) | 3 (3) | 10 (10)
DIARRHOEA (Gastrointestinal disorders) | 60 (84) | 63 (87) | 18 (26) | 12 (14)
NAUSEA (Gastrointestinal disorders) | 19 (20) | 27 (31) | 8 (9) | 11 (11)
VOMITING (Gastrointestinal disorders) | 18 (18) | 8 (9) | 5 (6) | 5 (5)
NASOPHARYNGITIS (Infections and infestations) | 22 (29) | 28 (34) | 6 (7) | 11 (14)
URINARY TRACT INFECTION BACTERIAL (Infections and infestations) | 18 (23) | 14 (19) | 6 (6) | 6 (6)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 22 (27) | 22 (23) | 8 (10) | 5 (6)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 16 (18) | 13 (15) | 4 (7) | 5 (7)
BLOOD PRESSURE INCREASED (Investigations) | 17 (18) | 16 (23) | 4 (4) | 5 (5)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 18 (19) | 8 (8) | 2 (3) | 2 (2)
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 16 (18) | 8 (9) | 6 (6) | 12 (13)
HEADACHE (Nervous system disorders) | 15 (20) | 20 (29) | 7 (7) | 12 (12)
HYPERTENSION (Vascular disorders) | 59 (72) | 58 (76) | 11 (13) | 12 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No